CLINICAL TRIAL: NCT03320369
Title: Effect of Elemental Diet on Adult Patients With Eosinophilic Gastroenteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-2766; U54AI117804 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-09

CONDITIONS: Eosinophilic Gastroenteritis
MeSH Terms: conditions — Eosinophilic enteropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): Elemental formula Intervention: Elemental Diet Therapy
  Interventions: Other: Elemental Diet Therapy

INTERVENTIONS:
Other: Elemental Diet Therapy — Elemental diet is a formula composed of amino-acids, carbohydrates, and lipids that is 100% nutritionally complete

SUMMARY:
The purpose of this study is to investigate the effect of an elemental diet on adult patients with Eosinophilic Gastroenteritis

DETAILED DESCRIPTION:
This prospective interventional study will investigate the effect of an exclusive, six week elemental diet in adult patients with Eosinophilic Gastroenteritis

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand and provide informed consent
2. Males and Females ≥18 to 65 years of age;
3. Have diagnosis of EG/EGE
4. Have histologically confirmed active disease > 30 eosinophils/hpf
5. Symptomatic (have experienced symptoms within the last one months prior to enrollment).
6. Female subjects of childbearing potential must have a negative pregnancy test upon study entry
7. Female (and male) subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study-specific methods may be listed, if applicable

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Secondary causes of gastrointestinal and peripheral eosinophilia
3. Eosinophilic infiltration isolated to the esophagus.
4. Pregnancy
5. Immunodeficiency states
6. Have been treated with topical swallowed steroids within the last 6 weeks or systemic steroids within the last 2 months unless repeat endoscopy is performed and shows active inflammation on these therapies in which case these medications will be allowed to be continued without dose escalation.
7. Have taken immunosuppression medication or immunomodulators within 2 months of the study unless the recent/baseline endoscopy has active histologic inflammation while on these medications. In this case, these medications will be permitted to be continued as long as the dose is not escalated during the treatment phase.
8. Have been on an elemental diet previously for six weeks with follow up endoscopy completed.
9. Have participated in any investigative drug study within 6 weeks prior to study entry.
10. Unable to complete study procedures including endoscopy.
11. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala Gonsalves, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gonsalves N, Doerfler B, Zalewski A, Yang GY, Martin LJ, Zhang X, Shoda T, Brusilovsky M, Aceves S, Thompson K, Rudman Spergel AK, Furuta G, Rothenberg ME, Hirano I. Prospective study of an amino acid-based elemental diet in an eosinophilic gastritis and gastroenteritis nutrition trial. J Allergy Clin Immunol. 2023 Sep;152(3):676-688. doi: 10.1016/j.jaci.2023.05.024. Epub 2023 Jul 18. PMID 37462600
- See also: Related info — http://www.rarediseasesnetwork.org/cms/CEGIR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants in Complete Histologic Remission
Description: Percent of patients who have achieved complete histologic remission. Complete histologic remission is defined as normalization of gastric mucosal eosinophilia (histology with less than the diagnostic threshold levels of mucosal eosinophilia (<30 eosinophils per high power field (HPF))
Time Frame: 6 weeks after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 15
percentage of participants | 100 [78 to 100]

2. Secondary Outcome: Percent of Participants in Partial Histologic Remission
Description: Percent of participants in partial histologic remission. Partial remission is defined as 50% or more reduction in the maximum of gastric and duodenal peak eosinophil count.
Time Frame: 6 weeks after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 15
percentage of participants | 93 [68 to 100]

3. Secondary Outcome: Mean Change From Baseline in Maximum Eosinophil Count
Description: The maximum between gastric and duodenal eosinophil counts per high power field were obtained at baseline and 6 weeks. Mean change in count is defined as maximum eosinophil count per high power field (hpf) at 6 weeks minus maximum eosinophil count per hpf at baseline. A reduction (negative change from baseline) in eosinophil count per hpf indicates improvement. Eosinophil counts per hpf from gastric and duodenal biopsies were assessed by research pathologists at 400X magnification.
Time Frame: Baseline, 6 weeks after treatment
Measure: Mean (95% Confidence Interval); unit: eosinophil counts per high power field
Arm/Group | Treatment
Number analyzed (Participants) | 15
eosinophil counts per high power field
  Baseline | 63.1 [50.6 to 75.5]
  Change | -46.9 [-59.1 to -34.7]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Total Gastric Endoscopic Reference Score
Description: The gastric endoscopic reference score utilizes standardized criteria for the presence and degree of major endoscopic features. Overall scores range from 0 - 10. Endoscopic features were assessed at baseline and 6 weeks. Change in overall endoscopic reference score is defined as overall score at 6 weeks minus overall score at baseline. A reduction (negative change) in score indicates improvement.
Time Frame: Baseline, 6 weeks after treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale
  Baseline Endoscopic Score | 5 [4 to 5]
  Change in Endoscopic Score | -3 [-3 to -2]

5. Secondary Outcome: Change From Baseline in Symptoms of Dyspepsia (SODA)
Description: The SODA questionnaire captures symptoms associated with gastric dyspepsia including symptoms associated with "pain" and "non-pain" as well as general satisfaction with present symptoms. The scores range from 0 to 47 for pain; 0 to 35 for non-pain, and 0 to 23 for satisfaction. Higher scores indicate more frequent and/or severe symptoms for pain and non-pain. Higher scores indicate greater satisfaction. Scores were obtained at baseline and 6 weeks. Change in score is defined as total score at 6 weeks minus total score at baseline. A reduction (negative change) indicates improvement in pain and non-pain. An increase (positive change) indicates improvement in satisfaction.
Time Frame: Baseline, 6 weeks after treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale
  Baseline Pain | 21.8 [16.1 to 27.5]
  Baseline Non Pain | 15.7 [13.8 to 17.7]
  Baseline Satisfaction | 9.2 [6.1 to 12.3]
  Change in Pain | -6.9 [-11.3 to -2.6]
  Change in Non Pain | -1.6 [-3.1 to -0.1]
  Change in Satisfaction | 6.1 [3.7 to 8.6]

6. Secondary Outcome: Change From Baseline in Promis Anxiety
Description: The Promis 29 questionnaire was used to assess anxiety. The range of scores for the anxiety sub-domain is 4 - 20 (raw score) with T-scores ranging from 40 to 82. A higher T-score indicates greater anxiety. Scores were obtained at baseline and 6 weeks. Change in score is defined as total score at 6 weeks minus total score at baseline.
Time Frame: Baseline, 6 weeks after treatment
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Treatment
Number analyzed (Participants) | 15
T-score
  Baseline Anxiety | 52.6 [47.2 to 58.0]
  Change in Anxiety | -2.7 [-7.0 to 1.6]

ADVERSE EVENTS:
Time Frame: From informed consent to cessation of treatment which is approximately 8 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=18)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=18)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Common Cold (General disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03320369/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03320369/SAP_001.pdf